CLINICAL TRIAL: NCT06816394
Title: Tarlatamab for Patients With Previously Treated Advanced Extrapulmonary Small Cell Carcinoma and Neuroendocrine Carcinoma
Brief Title: Tarlatamab for Advanced Extrapulmonary Small Cell Carcinoma and Neuroendocrine Carcinoma (TAURUS)
Acronym: TAURUS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202412002MIFE; 20247089 (Other Grant/Funding Number: Amgen)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Extrapulmonary Small Cell Carcinoma and Neuroendocrine Carcinoma
Keywords: tarlatamab; extrapulmonary small cell carcinoma; neuroendocrine carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tarlatamab (Experimental)
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — All subjects will receive a step dose (1 mg tarlatamab) on cycle 1 day 1 administered as a 60-minute intravenous (IV) infusion then 10 mg tarlatamab IV administered on cycle 1 day 8, cycle 1 day 15, and every 2 weeks (Q2W) thereafter.

SUMMARY:
Extrapulmonary small cell carcinoma (EPSCC) or neuroendocrine carcinoma (NEC) is a rare but fatal disease. The prognosis of patients with advanced EPSCC or NEC failed platinum-etoposide chemotherapy is poor with median overall survival ranged 6 to 9 months. High expression levels of DLL3 has been demonstrated in many EPSCC or NEC. As tarlatamab, a bispecific T-cell engager with dual affinity for DLL3 on tumor cells and CD3 on T cells, has demonstrated clinically meaningful activity for patients with advanced small cell lung cancer. We thus hypothesize that tarlatamab also has clinically activity for patients with advanced EPSCC and NECs.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Failed prior platinum-based chemotherapy
3. Histologically proven extrapulmonary small cell carcinoma or neuroendocrine carcinoma from gastrointestinal tract, genitourinary tract, gynecologic origin, and head and neck or unknown primary. When mixed histology (ex, adenocarcinoma, squamous cell carcinoma or transitional carcinoma) is found, small cell carcinoma or neuroendocrine carcinoma should be the predominant part.
4. Measurable lesions by RECIST 1.1 within 28 days prior to the first dose of tarlatamab.
5. ECOG Performance Status (PS) of 0 or 1.
6. Age greater or equal to 18 years old.
7. Subjects willing to provide archived tumor tissue samples (formalin fixed, paraffin embedded [FFPE] sample) or willing to undergo pretreatment tumor biopsy.
8. Subjects with treated brain metastases are eligible provided they meet the following criteria:

   1. Definitive therapy was completed at least 2 weeks prior to the first dose of tarlatamab.
   2. There is no evidence of radiographic central nervous system (CNS) progression following definitive therapy and by the time of study screening.
   3. Any CNS disease is asymptomatic for at least 7 days (unless symptoms are deemed irreversible by the investigator), the patient is off steroids for at least 7 days (physiologic doses of steroids are permitted), and the subject is off or on stable doses of anti-epileptic drugs for malignant CNS disease for at least 7 days.
9. Adequate organ function, defined as follows:

   1. hematological function:

      1. absolute neutrophil count ≥ 1.5 x 109/L
      2. platelet count ≥ 100 x 109/L
      3. hemoglobin > 9 g/dL (90 g/L)
   2. coagulation function:

      (1) prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) or activated partial thromboplastin time (APTT) ≤ 1.5 x institutional upper limit of normal (ULN). Subjects on chronic anticoagulation therapy who do not meet the criteria above may be eligible to enroll after discussion with the chief investigator.
   3. renal function:

      (1) estimated glomerular filtration rate (eGFR) based on Modification of Diet in Renal Disease (MDRD) calculation > 30 mL/min/1.73 m2.
   4. hepatic function:

      1. aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) < 3 x ULN (or < 5 x ULN for subjects with liver involvement).
      2. total bilirubin < 1.5 x ULN (or < 2 x ULN for subjects with liver metastases).
   5. pulmonary function:

      1. no clinically significant pleural effusion
      2. baseline oxygen saturation > 90% on room air
   6. cardiac function: (1) cardiac ejection fraction ≥ 50%, no clinically significant pericardial effusion as determined by an echocardiogram (ECHO) and no clinically significant electrocardiogram (ECG) findings

Exclusion Criteria:

1. Uncontrolled brain metastasis and leptomeningeal disease.
2. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
3. Prior exposure to DLL3 targeting agent.
4. Subjects who experienced recurrent pneumonitis (grade 2 or higher) or severe, life-threatening immune-mediated adverse events or infusion-related reactions including those that lead to permanent discontinuation while on treatment with immuno-oncology agents.
5. Unresolved toxicity from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1, or to levels dictated in the eligibility criteria with the exception of alopecia or toxicities from prior anti-tumor therapy that are considered irreversible (defined as having been present and stable for > 21 day) which may be allowed.
6. History of other malignancy within the past 2 years, with the following exceptions:

   1. malignancy treated with curative intent and with no known active disease present for > 2 years before enrollment and felt to be at low risk for recurrence by the treating physician.
   2. adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. adequately treated cervical carcinoma in situ without evidence of disease.
   4. adequately treated breast ductal carcinoma in situ without evidence of disease.
   5. prostatic intraepithelial neoplasia without evidence of prostate cancer.
   6. adequately treated urothelial papillary non-invasive carcinoma or carcinoma in situ.
7. Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months of first dose of tarlatamab.
8. History of arterial thrombosis (e.g., stroke or transient ischemic attack) within 12 months of first dose of tarlatamab.
9. Presence of fungal, bacterial, viral, or other infection requiring oral or IV antimicrobials for management within 7 days of first dose of tarlatamab with the exception:

   a. Those who have an active infection requiring parenteral antibiotic treatment: simple urinary tract infection and uncomplicated bacterial pharyngitis are permitted if responding to active treatment. Subjects requiring oral antibiotics who have been afebrile for >24 hours, have no leukocytosis, nor clinical signs of infection are eligible.
10. History of hypophysitis or pituitary dysfunction.
11. Exclusion of hepatitis infection based on the following results and/or criteria:

    1. Active hepatitis C infection (subjects with detectable hepatitis C antibody [HCV Ab] and HCV RNA viral load above the limit of quantification)

       (1) Subjects with presence of HCV Ab and HCV RNA viral load below the limit of quantification (HCV RNA negative) with or without prior treatment are allowed.
    2. Active hepatitis B infection (presence of hepatitis B surface antigen [HBsAg] and hepatitis B virus [HBV] DNA viral load above the limit of quantification [HBV DNA positive])

       1. Subjects with resolved HBV infection defined as absence of HBsAg and presence of HBV core antibody (anti-HBc) followed by an HBV DNA viral load below the limit of quantification (HBV DNA negative) are allowed, with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines.
       2. Subjects with chronic HBV infection inactive carrier state defined as presence of HBsAg and HBV DNA viral load below the limit of quantification [HBV DNA negative] are allowed, with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines.
12. Major surgery within 28 days of first dose tarlatamab.
13. Subject received prior therapy with tarlatamab.
14. Prior anti-cancer therapy within 30 days prior to first dose of tarlatamab.

    Exceptions:
    1. Subjects who received conventional chemotherapy are eligible if at least 14 days have elapsed and if all treatment-related toxicity has been resolved to grade ≤ 1.
    2. Prior palliative radiotherapy must have been completed at least 7 days before the first dose of tarlatamab.
15. Subjects has a diagnosis of immunodeficiency (e.g., positive/non-negative test for human immunodeficiency virus) except subjects on antiviral therapy and undetectable viral load are permitted with a requirement for regular monitoring for reactivation for the duration of treatment on study per local or institutional guidelines or subject is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of tarlatamab.
16. The following vaccines (live and live-attenuated vaccines) are excluded during the following study periods:

    1. Screening and during study treatment: live and live-attenuated vaccines are prohibited within 28 days prior to the first dose of tarlatamab and for the duration of the study.

       (1) Live viral non-replicating vaccine (e.g., Jynneos) for Monkeypox infection is allowed during the study (except during cycle 1) in accordance with local standard of care and institutional guidelines.
    2. End of study treatment: live and live-attenuated vaccines can be used when at least 60 days (5 x half-life of tarlatamab) have passed after the last dose of tarlatamab.
17. Subjects unwilling to use contraception or practice abstinence during treatment and for an additional 60 days after the last dose of tarlatamab.
18. Female subjects who are breastfeeding or who plan to breastfeed while on study through 60 days after the last dose of tarlatamab.
19. Male subjects unwilling to abstain from donating sperm during treatment and for an additional 60 days after the last dose of tarlatamab.
20. Female subjects planning to become pregnant while on study through 60 days after the last dose of tarlatamab.
21. Female subjects of childbearing potential with a positive pregnancy test assessed at screening and/or day 1 by a highly sensitive urine or serum pregnancy test.
22. Subject has known sensitivity to any of the products or components to be administered during dosing.
23. Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (e.g., Clinical Outcome Assessments) to the best of the subject and investigator's knowledge.
24. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) per RECIST 1.1 by investigator | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Please Select, Taiwan